CLINICAL TRIAL: NCT00823433
Title: Does Oral Penicillin Reach and Simulate Intravenous Penicillin Levels in Venous Umbilical Cord Blood of Laboring Pregnant Patients?
Brief Title: Oral Penicillin and Penicillin Levels in Venous Umbilical Cord Blood
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, John Uckele, Attending Physician, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008-183
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Group B Streptococcus
Keywords: Penicillin; Group B Streptococcus; Pregnancy; Labor
MeSH Terms: interventions — Penicillin V

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Penicillin (Experimental): 2 grams of oral penicillin V given within 4 hours of delivery
  Interventions: Drug: oral penicillin V

INTERVENTIONS:
Drug: oral penicillin V — 2 grams of oral penicillin V given within 4 hours of delivery.

SUMMARY:
Pregnant,laboring women will receive 2 grams of oral penicillin V before delivery. At the time of delivery of the infant, umbilical vein cord blood will be obtained from the umbilical cord. These cord blood samples will be sent for bioassay of penicillin levels.

DETAILED DESCRIPTION:
According to the CDC, before screening for GBS colonization was implemented, early onset GBS disease occurred at a rate of 1.5-2 per 1,000 live births. Antibiotic treatment for GBS colonized women according to guideline recommended by the American College of Obstetricians and Gynecologists (ACOG) decreases the risk for early onset neonatal GBS infection 10 fold. Unfortunately, many eligible women don't receive the full treatment protocol. Although the rate of early onset infection is low, the newborns of group B strep positive women who do not receive the recommended preventative antibiotics must undergo testing and extended observation.

This study will determine the level of antibiotics in the umbilical vein cord blood of newborn infants after the administration of penicillin orally while in labor and compare these levels to levels of penicillin in the umbilical vein cord blood of patients treated with intravenous penicillin in labor. Comparisons will be done through literature only; there will be no intravenous penicillin administration arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women admitted for delivery or for induction of labor
* singleton pregnancy
* 18 years old or older
* beyond 36 weeks gestation
* able to comprehend study and give informed consent

Exclusion Criteria:

* known history of beta-lactam antibiotic allergy
* impaired renal function
* multiple gestation
* current use of antibiotics
* plan to bank cord blood after delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The level of antibiotics in the umbilical vein cord blood of newborn infants after the administration of penicillin orally while in labor. | after delivery

SECONDARY OUTCOMES:
Compare levels of penicillin in the umbilical cord blood of women who received oral penicillin to the levels of women who received intravenous penicillin in labor. Comparisons will be done through literature only. | after delivery

CONTACTS AND LOCATIONS:
Overall Officials: John E Uckele, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States